CLINICAL TRIAL: NCT00223223
Title: Levetiracetam for Neuroprotection Against Corticosteroid-induced Hippocampal Dysfunction: A Proof of Concept Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: E. Sherwood Brown PI, UT Southwestern Medical Center at Dallas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 112004-003
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2005-09

CONDITIONS: Memory Loss Associated With Corticosteroid Use; Manic State Associated With Corticosteroid Use
MeSH Terms: interventions — Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam, Keppra

SUMMARY:
The purpose of this research is to determine whether the memory impairment and manic symptoms (feelings of agitation, overexcitement or hyperactivity) typically seen in those on corticosteroid therapy is decreased with a seizure medication called levetiracetam compared to placebo (an inactive substance). Since increased levels of cortisol (the body's natural corticosteroid) in the body are frequently associated with memory impairment interventions that may prevent or reverse this are of great importance.

It is hypothesized that patients who are scheduled to receive prescription corticosteroid therapy who are given levetiracetam pretreatment will show lesser memory impairment and manic symptoms than those receiving placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* Scheduled to receive a corticosteroid "burst" of at least 10 mg of prednisone equivalents and for at least 5 days duration
* English- or Spanish-speaking

Exclusion Criteria:

* History of allergic reaction or other contraindication to levetiracetam therapy
* Other unstable medical conditions (e.g. recent myocardial infarction, renal failure, diabetes with poor glycemic control)
* Pregnant or nursing women
* History of mental retardation, dementia or other severe cognitive disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-02; Primary Completion 2005-11 (Actual); Study Completion 2005-11

CONTACTS AND LOCATIONS:
Overall Officials: E. Sherwood Brown, M.D., Ph.D., Principal Investigator — UT Southwestern Medical Center at Dallas
Locations (1):
- The University of Texas Southwestern Medical Center, Dallas, Texas, United States